CLINICAL TRIAL: NCT07045441
Title: Patient Adherence to Splint Therapy and Counseling Programs in Temporomandibular Disorders: Development and Validation of a New Questionnaire
Brief Title: Development and Validation of a Temporomandibular Disorders (TMDs) Adherence Questionnaire
Acronym: TMDs
Status: Completed | Type: Observational
Sponsor: Soaad Tolba Mohammed Tolba Badawi (Other)
Responsible Party: Sponsor-Investigator, Soaad Tolba Mohammed Tolba Badawi, Lecturer of Oral and Maxillofacial Surgery, Faculty of Dentistry, Mansoura University, Egypt, Mansoura University
Organization: Mansoura University (Other)
Other Study IDs: RP.25.05.2
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Temporomandibular Disorders (TMDs); Splint Therapy; Behavioral Counseling; Treatment Adherence and Compliance
Keywords: Temporomandibular joint disorder; TMD adherence; Splint compliance; Counseling adherence; Psychometric validation; Questionnaire development; Conservative TMD treatment
MeSH Terms: conditions — Temporomandibular Joint Disorders; Treatment Adherence and Compliance | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TMD Patients Receiving Conservative Treatment: This cohort includes patients diagnosed with TMDs who received conservative treatment (splint therapy and behavioral counseling) for at least 6 months prior to participation. Adherence data were collected retrospectively through a structured questionnaire.
  Interventions: Other: Conservative Management for TMD

INTERVENTIONS:
Other: Conservative Management for TMD — This intervention includes a standardized conservative treatment protocol for TMDs, comprising splint therapy and a structured counseling program. The counseling covers education on diagnosis, medication adherence, dietary modifications, posture and behavior correction, sleep hygiene, parafunctional habit avoidance, physiotherapy exercises, pain and stress management, and importance of follow-up visits. Patients receive individualized instructions and monitoring as part of their routine clinical care. Adherence to these components is measured after 6 months of treatment using a validated adherence questionnaire.

SUMMARY:
The goal of this observational study is to assess patient adherence to splint therapy and behavioral counseling among individuals diagnosed with TMDs. The study uses a newly developed bilingual (Arabic and English) questionnaire to evaluate adherence behaviors. The main question it aims to answer is:

How consistently do TMDs patients follow conservative treatment protocols, including splint use and counseling recommendations?

Participants who are already receiving splint therapy and counseling as part of their standard care will complete the questionnaire to help researchers validate the tool and understand adherence patterns.

Last updated on June 20, 2025.

DETAILED DESCRIPTION:
This observational study aims to validate a newly developed adherence questionnaire tailored to measure patient compliance with conservative treatment protocols of TMDs, including splint therapy and behavioral counseling. The questionnaire was developed in both Arabic and English and underwent content validation, pilot testing, and psychometric evaluation.

Participants included in the study are individuals already undergoing treatment for TMD, specifically splint therapy and counseling, as part of their standard clinical care. The study does not assign any interventions but focuses on collecting data through patient-reported responses to the adherence questionnaire.

Data collected will be used to assess the questionnaire's reliability, validity, and factor structure to establish it as a robust tool for clinical and research settings. The outcomes of this study are expected to support the identification of non-adherent patients and facilitate targeted interventions to enhance treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Diagnosed with TMDs based on DC/TMD criteria
* Completed at least 6 months of conservative treatment (e.g., splint therapy and counseling program)
* Able to read and understand Arabic or English
* Provided informed consent

Exclusion Criteria:

* History of Temporomandibular joint (TMJ) surgery
* Currently undergoing other TMD-related treatments
* Presence of systemic musculoskeletal disorders (e.g., fibromyalgia, rheumatoid arthritis)
* Cognitive or psychiatric disorders impairing ability to participate
* Incomplete treatment duration (less than 6 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with TMDs who have completed six months of conservative treatment, including splint therapy and behavioral counseling.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Content Validity of the Adherence Questionnaire | Preceding patient data collection (before pilot phase)
  Assessment of content validity using expert panel ratings to compute Item Content Validity Index (I-CVI) and Content Validity Ratio (CVR).
  Unit of Measure: I-CVI and CVR values
Internal Consistency of the Adherence Questionnaire | Baseline (after 6 months of treatment)
  Evaluation of the internal consistency of the items of adherence questionnaire using Cronbach's alpha across all domains and total score. Unit of Measure: Cronbach's alpha coefficient

SECONDARY OUTCOMES:
Test-Retest Reliability of the Adherence Questionnaire | 1-week interval after baseline administration
  Assessment of temporal stability using Intraclass Correlation Coefficient (ICC) between two administrations of the questionnaire, 1 week apart.
  Unit of Measure: ICC
Construct Validity via Exploratory Factor Analysis (EFA) | Baseline (after 6 months of treatment)
  Evaluation of construct validity through Exploratory Factor Analysis to identify the underlying factor structure.
  Unit of Measure: Number of factors extracted and percent variance explained

CONTACTS AND LOCATIONS:
Overall Officials: Soaad Tolba Badawy, Lecturer, Oral Surgery, MU, Principal Investigator — Faculty of dentistry, Mansoura university
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The decision regarding sharing of individual participant data (IPD) has not yet been finalized. Further details will be provided when available

REFERENCES:
- [Derived] Badawy ST, Badawi AT, Haggag MA. Patient Adherence to Splint Therapy and Counselling Programmes in Temporomandibular Disorders: Development and Validation of a New Questionnaire. J Oral Rehabil. 2026 Jan 24. doi: 10.1111/joor.70153. Online ahead of print. PMID 41578714